CLINICAL TRIAL: NCT02388113
Title: The Effect of Accumulated Versus Traditional Exercise Training on Metabolic Control and Heart Function in Individuals With Type 2 Diabetes
Brief Title: Effect of Exercise Frequency on Metabolic Control and Heart Function in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1405
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise therapy; Time factors
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- accumulated exercise (Experimental): 12 exercise sessions of 10 minutes each week, 2 per day, 1 day rest
  Interventions: Behavioral: accumulated exercise
- traditional exercise (Active Comparator): 4 exercise sessions of 30 minutes each week, 3 in the training laboratory, 1 at home.
  Interventions: Behavioral: traditional exercise

INTERVENTIONS:
Behavioral: accumulated exercise
  Arms: accumulated exercise
Behavioral: traditional exercise
  Arms: traditional exercise

SUMMARY:
This study will compare two interventions with the same exercise intensities and caloric expenditure but with different exercise frequency, on metabolic control and other risk factors in individuals with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes

Exclusion Criteria:

* insulin treatment
* severe chronic diabetic complications
* liver dysfunction
* kidney dysfunction
* inflammatory diseases
* heart failure
* myocardial ischemia
* major cardiovascular event history
* physical exercise more than current guidelines for type 2 diabetes
* inability to exercise

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
glycosylated hemoglobin (HbA1c) | 12 weeks
  The measured HbA1c level consists of average blood glucose by 50% from the last month, 25% from the previous month, and 25% by the two first previous months. Analysis: standard procedure of St Olavs Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Ingul, PhD MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Diagnostic Imaging, Trondheim, Norway